CLINICAL TRIAL: NCT00405288
Title: The Safety of Proctofoam-HC in the Third Trimester of Pregnancy
Status: Completed | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Duchesnay Inc. (Industry)
Responsible Party: Principal Investigator, Gideon Koren, Chief, Global Child Health, The Hospital for Sick Children
Other Study IDs: 1000008482
Record Dates: First submitted 2006-11-28; First posted 2006-11-30 (Estimated); Results first posted 2014-02-05 (Estimated); Last update posted 2014-02-05 (Estimated); Status verified 2014-01

CONDITIONS: Hemorrhoids; Pregnancy
Keywords: Hemorrhoids; Pregnancy; antihemorrhoidal; Proctofoam; infants
MeSH Terms: conditions — Hemorrhoids | interventions — proctofoam-HC

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Proctofoam-HC®: Women in the third trimester of pregnancy prescribed Proctofoam-HC® aerosol foam canister for 36 applications for treatment of symptoms of hemorrhoids. One applicatorful is to be applied into the anus (or on the perianal area) two or three times daily and after bowel evacuation.
  Interventions: Drug: Proctofoam-HC®
- Control: Control group of women in the third trimester of pregnancy who were not exposed to any teratogens during the course of the pregnancy, and to Proctofoam-HC any of its components, or any other topical corticosteroids or local anaesthetics during the course of their pregnancy.

INTERVENTIONS:
Drug: Proctofoam-HC® — Observational study of the exposure to Proctofoam-HC®
  Other Names: 1% Pramoxine+1% Hydrocortisone ( Proctofoam-HC®)
  Groups: Proctofoam-HC®

SUMMARY:
The purpose of this study is to evaluate the fetal safety of topical application of Proctofoam-HC®, an antihemorrhoidal, in the third trimester of pregnancy.

DETAILED DESCRIPTION:
Hemorrhoids are a frequent condition in pregnancy. The rate is increased as pregnancy progresses, and they affect up to 24% of pregnant women in the third trimester. Complications of untreated hemorrhoids include bleeding, prolapse, soiling, discharge with perianal irritation and itching, and in severe cases, severe pain and venous engorgement which could even lead to thrombosis and infarction. Hemorrhoids are treated with a variety of suppositories and gels, based on analgesic and anti-inflammatory effects. The safety of these antihemorrhoidal products has not yet been documented in pregnant women.

Proctofoam-HC® has been on the Canadian market for 25 years. It combines the anti-inflammatory action of hydrocortisone with the surface anesthetic effect of pramoxine HCl. It is approved for temporary relief of anorectal inflammation, pruritus, pain and swelling associated with haemorrhoids, fissures, pruritus ani, cryptitis, proctitis and postoperative pain.

We hypothesize that local application of Proctofoam-HC® in the third trimester of pregnancy is safe for the mother and fetus.

ELIGIBILITY:
Inclusion Criteria:

* For intervention group, any pregnant woman with a primary anorectal condition during the third trimester of pregnancy
* For control group, women in third trimester of pregnancy not treated with Proctofoam, and matched on maternal age and smoking status
* for either group,no other pregnancy complications

Exclusion Criteria:

* exposure to known teratogens during pregnancy as evident either during the prenatal or postnatal interview
* insufficient English language skills to understand the questionnaires and assessment material
* Women who have received other corticosteroid medications (systemic or topical)during pregnancy
* Women with the following conditions: abscess, fistula, tuberculosis, varicella, acute Herpes Simplex or fungal infection
* age less than 18 years
* History of previous reaction to any of the product's components, such as: local irritation, hypertrichosis, hypopigmentation, etc.
* Known Intrauterine Growth Restriction (IUGR) or a chronic state that may cause IUGR (SLE, placental insufficiency).
* Multi fetal pregnancy
* Binge alcohol consumption (5 or more drinks on one occasion,in a row or within a short period of time)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant woman with a primary anorectal condition during the third trimester of pregnancy and pregnant women in the third trimester of pregnancy without anorectal condition
Sampling Method: Probability Sample
Enrollment: 408 (Actual)
Dates: Start 2006-11; Primary Completion 2009-11 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gideon Koren, MD, Principal Investigator — The Hospital for Sick Children, Toronto Canada
Locations (2):
- Canada (2):
  - Mount Sinai Hospital, Toronto, Ontario
  - The Hospital for Sick Children, Toronto, Ontario

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In this multicentre study we recruited pregnant women who were prescribed Proctofoam-HC for hemorrhoids by their physicians and who completed two telephone interviews using two specially designed questionnaires.
Pre-assignment Details: There were no significant events that occur before assignment of the enrolled patients to groups.
Groups:
- Proctofoam-HC®: Proctofoam-HC® aerosol foam canister for 36 applications. One applicatorful should be injected into the anus (or perianal area) two or three times daily and after bowel evacuation.
- Control: Control, who were not exposed to any teratogens during the course of the pregnancy and to Proctofoam-HC, any of its components, or any other topical corticosteroids or local anaesthetics during the course of their pregnancy.
Period: Overall Study
Arm/Group | Proctofoam-HC® | Control
Started | 204 | 204
Completed | 204 | 204
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Proctofoam-HC® | Control | Total
Number analyzed (Participants) | 204 | 204 | 408
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 204 | 204 | 408
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32 (4.9) | 31.5 (4.9) | 31.75 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 204 | 204 | 408
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 204 | 204 | 408

OUTCOME MEASURES:

1. Primary Outcome: Birth-weight
Description: Weight of the baby measured in grams at time of birth.
Time Frame: until delivery
Population: Estimated number of 200 patients per arm, to detect significant difference of 200g in birth weight at a power of 80% and alpha of 5%. Seven pairs of twin pregnancies were excluded from the comparison of birth weight.
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Proctofoam-HC® | Control
Number analyzed (Participants) | 201 | 201
grams | 3406.9 (452.7) | 3487.7 (491.4)
Statistical Analysis 1: Comparison: Proctofoam-HC® vs Control; Null hypothesis: Birth weight in pregnancies exposed to Proctofoam-HC will be the same as control pregnancies. To detect a clinically significant decrease of 200 g in birth weight at a power of 80% and alpha of 5%, 200 women per group were required. Post hoc power analysis of our cohort revealed that, in fact, we had a 91.5% power to detect a 200 g difference in birth weight between the two groups; Test type: Superiority or Other; p = 0.17, t-test, 2 sided; Mean Difference (Final Values) = 50, 95% CI 2-sided [0 to 200], Standard Deviation 450

2. Secondary Outcome: Gestational Age at Delivery
Description: Fetal gestational age at delivery
Time Frame: until delivery
Measure: Mean (Standard Deviation); unit: gestational weeks
Arm/Group | Proctofoam-HC® | Control
Number analyzed (Participants) | 204 | 194
gestational weeks | 39.4 (1.4) | 39.1 (2.5)
Statistical Analysis 1: Comparison: Proctofoam-HC® vs Control; Test type: Superiority or Other; p = 0.16, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 1, 95% CI 2-sided [0 to 3], Standard Deviation 3

3. Secondary Outcome: Mode of Delivery
Description: Method of delivery for both groups: vaginal or caesarean section
Time Frame: at birth
Measure: Number; unit: participants
Arm/Group | Proctofoam-HC® | Control
Number analyzed (Participants) | 204 | 204
participants
  Vaginal delivery | 173 | 146
  Caesarean section | 31 | 55
  Unknown | 0 | 3
Statistical Analysis 1: Comparison: Proctofoam-HC® vs Control; The null hypothesis is that the proportion of vaginal deliveries in the Proctofoam and Control groups will be the same (ie. there will not be a greater proportion of complicated deliveries in either group); Test type: Superiority or Other; p = 0.003, McNemar; chi square = 30

4. Secondary Outcome: Prematurity
Description: birth at <37 gestational weeks
Time Frame: at birth
Measure: Number; unit: participants
Arm/Group | Proctofoam-HC® | Control
Number analyzed (Participants) | 201 | 190
participants
  yes | 8 | 10
  no | 193 | 180
Statistical Analysis 1: Comparison: Proctofoam-HC® vs Control; The null hypothesis is that the proportion of pre-term births in the Proctofoam and Control groups will be the same; Test type: Superiority or Other; p = 0.55, McNemar; chi square = 5

5. Secondary Outcome: Fetal Distress
Description: Presence of fetal distress at birth: heart deceleration/acceleration, meconium/amniotic fluid
Time Frame: at birth
Measure: Number; unit: participants
Arm/Group | Proctofoam-HC® | Control
Number analyzed (Participants) | 199 | 173
participants
  Fetal distress | 36 | 31
  No fetal distress | 163 | 142
Statistical Analysis 1: Comparison: Proctofoam-HC® vs Control; Fetal Distress The null hypothesis is that the proportion of fetal distress in the Proctofoam and Control groups will be the same; Test type: Superiority or Other; p = 0.97, McNemar; chi square = 10

6. Secondary Outcome: Low Birth Weight at Birth
Description: Low birth weight (birth weights <2500 grams)
Time Frame: at birth
Population: Per protocol, the estimated number of 200 patients per arm, to detect significant difference of 200g in birth weight (primary outcome) for a power of 80% and alpha of 5% was used.
Measure: Number; unit: participants
Arm/Group | Proctofoam-HC® | Control
Number analyzed (Participants) | 200 | 201
participants
  Yes | 6 | 3
  No | 194 | 198
Statistical Analysis 1: Comparison: Proctofoam-HC® vs Control; Low birth weight <2,500g; The null hypothesis is that the proportion of low birth weight babies in the Proctofoam and Control groups will be the same; Test type: Superiority or Other; p = 0.31, McNemar; binary = 3

7. Secondary Outcome: Neonatal Health
Description: Neonatal health at birthyes=need for medical attention or intervention after birth, abnormalities detected, no= no need for medical attention, no abnormalities detected at birth
Time Frame: at birth
Measure: Number; unit: participants
Arm/Group | Proctofoam-HC® | Control
Number analyzed (Participants) | 199 | 199
participants
  Yes (present neonatal health concerns) | 28 | 24
  No (absent neonatal health concerns) | 171 | 154
Statistical Analysis 1: Comparison: Proctofoam-HC® vs Control; The null hypothesis is that the proportion of healthy babies (not requiring NICU (neonatal intensive care unit) or additional medical monitoring) will be the same between the Proctofoam and Control groups; Test type: Superiority or Other; p = 0.87, McNemar; chi square = 10

8. Post Hoc Outcome: Cardiovascular Neonatal Health Concerns in the First Two Weeks After Birth
Description: Assessment of neonate's morphology and function of cardiovascular system in the first two weeks after birth
Time Frame: neonatal period
Measure: Number; unit: participants
Arm/Group | Proctofoam-HC® | Control
Number analyzed (Participants) | 199 | 179
participants
  Cardiovascular anomalies | 2 | 0
  Heart murmur | 6 | 4
  Premature atrial contraction | 0 | 2
Statistical Analysis 1: Comparison: Proctofoam-HC® vs Control; Test type: Superiority or Other; p = 0.99, Fisher Exact; proportion = 4

9. Post Hoc Outcome: Respiratory Neonatal Health Concerns
Time Frame: neonatal period
Measure: Number; unit: participants
Arm/Group | Proctofoam-HC® | Control
Number analyzed (Participants) | 199 | 178
participants
  Pulmonary aspiration | 4 | 0
  Mild asthma | 2 | 2
  Tachypnea | 0 | 2
Statistical Analysis 1: Comparison: Proctofoam-HC® vs Control; Test type: Superiority or Other; p = 0.99, Fisher Exact; proportion = 3

10. Post Hoc Outcome: Neonatal Health Concerns-infections
Description: Infections occuring in the neonatal period
Time Frame: neonatal period
Measure: Number; unit: participants
Arm/Group | Proctofoam-HC® | Control
Number analyzed (Participants) | 199 | 178
participants
  Urinary tract infections | 2 | 0
  Streptococcus B infection | 0 | 2
  Pneumonia | 0 | 2
  Leucocytosis | 2 | 0
Statistical Analysis 1: Comparison: Proctofoam-HC® vs Control; Test type: Superiority or Other; p = 0.99, Fisher Exact; proportion = 2

11. Post Hoc Outcome: Skin Conditions in Neonatal Period
Time Frame: neonatal period
Measure: Number; unit: participants
Arm/Group | Proctofoam-HC® | Control
Number analyzed (Participants) | 199 | 178
participants
  Rash | 2 | 2
  Eczema | 0 | 2
  Acne | 0 | 2
Statistical Analysis 1: Comparison: Proctofoam-HC® vs Control; Test type: Superiority or Other; p = 0.35, Fisher Exact; proportions = 2

12. Post Hoc Outcome: Other Neonatal Health Concerns
Time Frame: neonatal period
Measure: Number; unit: participants
Arm/Group | Proctofoam-HC® | Control
Number analyzed (Participants) | 199 | 178
participants
  Conjuctivitis | 4 | 0
  Myopia | 0 | 2
  Colic | 0 | 4
  Milk allergy | 0 | 2
  Hypoglycemia | 4 | 0
  Poor feeding | 2 | 0
  Poor weight gain | 2 | 2
  Anemia | 0 | 2
  Renal calculi | 0 | 2

ADVERSE EVENTS:
Time Frame: The data was collected within the 4 year study period.
Arm/Group | Proctofoam-HC® | Control
Serious Adverse Events (participants affected / at risk) | 0/204 | 0/204
Other Adverse Events (participants affected / at risk) | 0/204 | 0/204

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes